CLINICAL TRIAL: NCT04403087
Title: Additive Effect of Trimebutine on the Development of Adverse Events Related to the Helicobacter Pylori Eradication Medications; an Open-label, Randomized Controlled Trial
Brief Title: Trimebutine on the Development of Adverse Events Related to the Helicobacter Pylori Eradication Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, Associate professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCSHPAE
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Trimebutine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimebutine add group (Experimental): Addition of Trimebutine on the Bismuth-containing quadruple regimen
  Interventions: Drug: Trimebutine 100 MG
- Control group (No Intervention): Bismuth-containing quadruple regimen

INTERVENTIONS:
Drug: Trimebutine 100 MG — Trimebutine 100mg three times a day
  Other Names: Polybutine (Samil Pharm.Co.,Ltd.)
  Arms: Trimebutine add group

SUMMARY:
Adverse events related to the eradication medication is one of the reason of lower eradication success in the H. pylori treatment. The aim of this study was to evaluate the additive effect of trimebutine for the development of adverse events related to the H. pylori eradication regimen.

DETAILED DESCRIPTION:
Adverse events related to the eradication medication is one of the reason of lower eradication success in the H. pylori treatment. The common adverse events related to the eradication medications area as follows; Abdomen discomfort, pain, nausea, vomiting, diarrhea, bloating, urticaria, dizziness, headache, etc,. Various methods have been tried to reduce or prevent the adverse events related to the eradication medications. However, there is no established methods to reduce or prevent these events.

The aim of this study was to evaluate the additive effect of trimebutine for the development of adverse events related to the H. pylori eradication regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent upper gastrointestinal endoscopy and were proven to have H. pylori infection either by using the rapid urease test, the 13 C-urea breath test (UBT), or histological examination.

Exclusion Criteria:

* Subjects who took medications as Proton pump inhibitor, Histamin-2 receptor antagonist and antibiotics,
* Subjects who underwent stomach resection
* Subjects less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Overall compliance of eradication medication | 2 weeks after prescription of eradication medication
  How much the enrolled subjects took prescribed eradication medication

SECONDARY OUTCOMES:
Adverse events related to eradication medication | 2 weeks and 6 weeks after prescription of eradication medication
  percentage of Adverse events related to eradication medication

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, MD, PHD, Principal Investigator — Hallym University
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No